CLINICAL TRIAL: NCT01065103
Title: Fractional Flow Reserve Stability Study of Non-culprit Vessels in Patients With ST Elevation Myocardial Infarction
Brief Title: Fractional Flow Reserve (FFR) Stability in Non-Culprit Vessels at ST Elevation Myocardial Infarction(STEMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Wood, MD, Principal Investigator, Cardiology Research UBC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H09-03435
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction
Keywords: STEMI; Primary angioplasty; Non-culprit vessel at STEMI; Fractional Flow Reserve; ST-elevation myocardial infarction; Fractional Flow Reserve in non-culprit vessel at STEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FFR measurement (Experimental)
  Interventions: Procedure: FFR (Fractional Flow Reserve)

INTERVENTIONS:
Procedure: FFR (Fractional Flow Reserve) — Single FFR measurement in non-culprit vessel

SUMMARY:
It has been shown that if it can be accomplished within a 90 minute "door to balloon" time, opening an artery in an acute heart attack situation (ST elevation myocardial infarction or STEMI) is best treated with balloon angioplasty and stenting (percutaneous coronary intervention or PCI). In these situations, there may be narrowings other than the one causing the heart attack (culprit) and studies have shown that delaying treatment of other narrowings for follow-up procedure is better than intervening at the time of the acute MI.

DETAILED DESCRIPTION:
Prompt, sustained and complete reperfusion of the myocardium supplied by the infarct related artery (IRA) remains the cornerstone of therapy for the treatment of ST segment elevation myocardial infarction (STEMI). Although reperfusion can be achieved using fibrinolytic agents, it is generally accepted that primary percutaneous coronary intervention (PPCI) is preferable, with the caveat that it be performed promptly by experienced personnel.

It has been observed that up to 74% of patients with STEMI have evidence of multi-vessel disease (MVD) during angiography. The presence of MVD is independently associated with worse clinical outcomes and the presence of MVD at the time of STEMI is predictive of the need for future revascularization within 1 year, with over half of these repeat procedures driven by the development of unstable coronary syndromes 8. However, retrospective analyses have determined that immediate intervention upon non-culprit vessels (NCV) in addition to the IRA is associated with worse clinical outcomes compared to a strategy of intervening upon the IRA alone. Furthermore, small studies have shown no increase in mortality associated with a strategy with delayed (7 day) intervention of NCV compared to a strategy of intervening on the IRA alone. Accordingly, it is considered inappropriate to intervene upon non-culprit arteries in the absence of demonstrable ischemia following successful revascularization of the IRA in the setting of STEMI 11 and the 2007 ACC/AHA STEMI guidelines give a Class IIb recommendation for delayed intervention upon a hemodynamically significant NCV >24 hours after the index STEMI.

However, the guidelines do not provide guidance regarding how to define hemodynamic significance of the NCV, nor do they speak to the exact timing of when NCV revascularization should be performed after the initial 24 hours. Indeed, this ambiguity is reflected in local practice within the Vancouver Coastal Health Authority (R. Boone, personal communication), with some interventional cardiologists performing NCV revascularization during the index hospitalization prior to patient discharge, while others bring patients back within 6-8 weeks of the index STEMI for a "staged", elective revascularization of the NCV. Finally, other cardiologists will defer NCV revascularization entirely in the absence of recurrent ischemia.

There remains significant doubt as to the most appropriate treatment strategy for the STEMI patient who is found to have MVD. Unfortunately, this clinical dilemma is made more difficult by the observation that the angiographic and clinical assessment of the NCV remains imprecise in the STEMI setting. It remains unclear whether or not traditional angiographic assessment of the NCV is reliable over time following an index myocardial infarction, or if it can be used to reliably guide decision making for revascularization of NCV in the setting of STEMI. In one study, only 10% of lesions judged by visual assessment of the coronary angiogram to require NCV PCI following STEMI, were noted to be angiographically significant by quantitative coronary angiography at the time of the index angiogram 12. Finally, prior studies have demonstrated that the severity of non culprit lesions were found to be significantly exaggerated using traditional angiography at the time of the index MI. A study of 548 patients with acute MI and MVD revealed that 21% of NCV lesions initially thought to be >50% at the time of the index MI were found to be <50% at the time of subsequent angiography. Accordingly, there is significant interest in finding alternate means of assessing clinically and angiographically significant lesions in the setting of both stable and unstable coronary syndromes.

Fractional flow reserve (FFR) is a simple, reliable and reproducible physiological index of lesion severity. It is defined as the ratio between coronary artery pressure distal to a stenosis and aortic root pressure, measured following maximal dilation of the distal coronary resistance vessels. FFR is a reliable index of maximal achievable coronary flow. An FFR of <0.8 identifies ischemia-causing coronary stenoses with >90% accuracy. Conversely, lesions deemed nonsignificant by FFR can be safely treated medically with an annual rate of death or myocardial infarction of <1%. Recently, an FFR guided strategy for elective PCI was found to be superior to a strategy of coronary intervention guided by angiography alone. FFR has also been found to be a reliable modality for the hemodynamic assessment of coronary lesions in the setting of acute myocardial infarction, with a similar correlation between FFR and percent diameter stenosis of coronary vessels in the acute infarct setting compared to FFR amongst matched controls undergoing elective PCI. Additionally, FFR correlates well with the identification of residual reversible perfusion abnormalities shortly following an index myocardial infarction (MI). However, it remains unknown if an abnormal FFR of a NCV remains stable following an acute STEMI.

We are proposing a study to determine the precision and stability of FFR as a measure of lesion severity in NCV in patients undergoing clinically indicated revascularization of the culprit vessel in the setting of STEMI. Our hypothesis is that FFR will remain stable over time within myocardium that is not subtended by the infarct related artery. We believe FFR can potentially serve as a reliable and safe angiographic tool to guide delayed revascularization decisions for non-culprit vessels amongst STEMI patients with MVD.

STUDY SCHEMA Following successful revascularization of the IRA, patients deemed to be appropriate for a delayed revascularization procedure on a NCV (ie not during the index hospitalization) will undergo FFR of the NCV during the index catheterization. Consent for the FFR will be obtained prior to successful revascularization of the IRA. Patients with NCV stenoses who are brought back for planned elective revascularization of the NCV lesion(s), according to usual clinical practice following revascularization of the culprit lesion, will undergo repeat FFR on the NCV prior to planned revascularization. Patients who are deemed appropriate to undergo intervention on the NCV during the index hospitalization for clinical reasons will not be eligible for inclusion in this analysis.

ENDPOINTS The primary endpoint of this study will be the comparison of initial and repeat FFR of a NCV amongst STEMI patients with MVD deemed appropriate for delayed revascularization of the NCV. This study will not stipulate the timing of NCV revascularization; this decision will be made by the treating interventional cardiologist. However it is expected that most patients will undergo NCV revascularization within 4 to 8 weeks following the index hospital stay. Patients who require in-hospital revascularization of the NCV during the index hospitalization will not be enrolled into this study. Secondary endpoints of the trial will be the comparison of baseline and repeat FFR with digital subtraction quantitative angiography of the NCV. Tertiary endpoints will be the evaluation of major adverse cardiac events amongst enrolled patients through to the repeat procedure.

CLINICAL IMPACT We believe that the results of this proposed study could result in significant changes in the management of STEMI. A potential finding that FFR is a durable method of assessing the severity of the NCV in the setting of STEMI could lead to a shift towards the use of this technology to guide decision making for revascularization in acute coronary syndromes, similar to the paradigm shift seen in elective PCI following the publication of the FAME trial. Furthermore, our study will expand upon our understanding of the angiographic behaviour of nonculprit vessels in the setting of STEMI, which may serve to change future recommendations regarding revascularization decisions amongst patients with MVD who present with acute myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

1. Any patient >18 years of age with an acute STEMI eligible for primary PCI
2. Readily identifiable culprit vessel and at least one other (non-culprit) vessel of a least >50% severity by traditional angiography
3. Deemed appropriate for a strategy of delayed revascularization of the NCV.

Exclusion Criteria:

1. Inability to provide informed consent
2. Cardiogenic shock or severe (Killip III) congestive heart failure
3. Hemodynamically significant ventricular arrhythmias
4. Severe recurrent clinically significant ischemia following successful PCI of the IRA
5. Thrombocytopenia (platelet count <100,000)
6. Severe anemia (HgB <100 g/L)
7. Major bleeding during hospitalization of the index STEMI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
FFR measurement | Baseline and repeated at 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

REFERENCES:
- [Background] Canadian Cardiovascular Society; American Academy of Family Physicians; American College of Cardiology; American Heart Association; Antman EM, Hand M, Armstrong PW, Bates ER, Green LA, Halasyamani LK, Hochman JS, Krumholz HM, Lamas GA, Mullany CJ, Pearle DL, Sloan MA, Smith SC Jr, Anbe DT, Kushner FG, Ornato JP, Pearle DL, Sloan MA, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA 2004 guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):210-47. doi: 10.1016/j.jacc.2007.10.001. No abstract available. PMID 18191746
- [Background] Keeley EC, Grines CL. Primary percutaneous coronary intervention for every patient with ST-segment elevation myocardial infarction: what stands in the way? Ann Intern Med. 2004 Aug 17;141(4):298-304. doi: 10.7326/0003-4819-141-4-200408170-00010. PMID 15313746
- [Background] Keeley EC, Grines CL. Should patients with acute myocardial infraction be transferred to a tertiary center for primary angioplasty or receive it at qualified hospitals in the community? The case for emergency transfer for primary percutaneous coronary intervention. Circulation. 2005 Nov 29;112(22):3520-32; discussion 3533. No abstract available. PMID 16320379
- [Background] Koyama Y, Hansen PS, Hanratty CG, Nelson GI, Rasmussen HH. Prevalence of coronary occlusion and outcome of an immediate invasive strategy in suspected acute myocardial infarction with and without ST-segment elevation. Am J Cardiol. 2002 Sep 15;90(6):579-84. doi: 10.1016/s0002-9149(02)02559-6. PMID 12231080
- [Background] Hanratty CG, Koyama Y, Rasmussen HH, Nelson GI, Hansen PS, Ward MR. Exaggeration of nonculprit stenosis severity during acute myocardial infarction: implications for immediate multivessel revascularization. J Am Coll Cardiol. 2002 Sep 4;40(5):911-6. doi: 10.1016/s0735-1097(02)02049-1. PMID 12225715
- [Background] Goldstein JA, Demetriou D, Grines CL, Pica M, Shoukfeh M, O'Neill WW. Multiple complex coronary plaques in patients with acute myocardial infarction. N Engl J Med. 2000 Sep 28;343(13):915-22. doi: 10.1056/NEJM200009283431303. PMID 11006367
- [Background] Corpus RA, House JA, Marso SP, Grantham JA, Huber KC Jr, Laster SB, Johnson WL, Daniels WC, Barth CW, Giorgi LV, Rutherford BD. Multivessel percutaneous coronary intervention in patients with multivessel disease and acute myocardial infarction. Am Heart J. 2004 Sep;148(3):493-500. doi: 10.1016/j.ahj.2004.03.051. PMID 15389238
- [Background] Glaser R, Selzer F, Faxon DP, Laskey WK, Cohen HA, Slater J, Detre KM, Wilensky RL. Clinical progression of incidental, asymptomatic lesions discovered during culprit vessel coronary intervention. Circulation. 2005 Jan 18;111(2):143-9. doi: 10.1161/01.CIR.0000150335.01285.12. Epub 2004 Dec 27. PMID 15623544
- [Background] Kong JA, Chou ET, Minutello RM, Wong SC, Hong MK. Safety of single versus multi-vessel angioplasty for patients with acute myocardial infarction and multi-vessel coronary artery disease: report from the New York State Angioplasty Registry. Coron Artery Dis. 2006 Feb;17(1):71-5. doi: 10.1097/00019501-200602000-00012. PMID 16374145
- [Background] Chen LY, Lennon RJ, Grantham JA, Berger PB, Mathew V, Singh M, Holmes DR Jr, Rihal CS. In-hospital and long-term outcomes of multivessel percutaneous coronary revascularization after acute myocardial infarction. Am J Cardiol. 2005 Feb 1;95(3):349-54. doi: 10.1016/j.amjcard.2004.09.032. PMID 15670543
- [Background] Patel MR, Dehmer GJ, Hirshfeld JW, Smith PK, Spertus JA; American College of Cardiology Foundation Appropriateness Criteria Task Force; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association for Thoracic Surgery; American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography; Heart Failure Society of America; Society of Cardiovascular Computed Tomography. ACCF/SCAI/STS/AATS/AHA/ASNC 2009 Appropriateness Criteria for Coronary Revascularization: a report by the American College of Cardiology Foundation Appropriateness Criteria Task Force, Society for Cardiovascular Angiography and Interventions, Society of Thoracic Surgeons, American Association for Thoracic Surgery, American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography, the Heart Failure Society of America, and the Society of Cardiovascular Computed Tomography. J Am Coll Cardiol. 2009 Feb 10;53(6):530-53. doi: 10.1016/j.jacc.2008.10.005. PMID 19195618
- [Background] Lemesle G, de Labriolle A, Bonello L, Torguson R, Kaneshige K, Xue Z, Suddath WO, Satler LF, Kent KM, Lindsay J, Pichard AD, Waksman R. Incidence, predictors, and outcome of new, subsequent lesions treated with percutaneous coronary intervention in patients presenting with myocardial infarction. Am J Cardiol. 2009 May 1;103(9):1189-95. doi: 10.1016/j.amjcard.2009.01.029. Epub 2009 Mar 13. PMID 19406257
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] De Bruyne B, Pijls NH, Bartunek J, Kulecki K, Bech JW, De Winter H, Van Crombrugge P, Heyndrickx GR, Wijns W. Fractional flow reserve in patients with prior myocardial infarction. Circulation. 2001 Jul 10;104(2):157-62. doi: 10.1161/01.cir.104.2.157. PMID 11447079
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660